## ISOMETRIC CORE MUSCLE ENDURANCE IN HEALTHY ACTIVE AND NON- ACTIVE WORKING AGE POPULATIONS Hanna Holmberg, Lynne E Gaskell

28.05.2018

## **Research Participant Consent Form**

**Title of Project:** "Are there any differences in isometric core muscle endurance between old and young working-age populations with and without lower back pain?"

| Ethics Ref No: | | | |
|---|---|---|---|
| Name of Researcher: | | | |
| <ul> <li>(Delete as appropriate)</li> <li>□ I confirm that I have read and understood the participant information sheet for the above study and what my contribution will be.</li> </ul> | Yes | No | |
| ☐ I have been given the opportunity to ask questions (face to face,via telephone and e-mail) | Yes | No | |
| ☐ I agree to take part in the study | Yes | No | NA |
| ☐ I understand that my participation is voluntary and that I can withdraw from the research at any time without giving any reason. If I decide to withdraw, the data I have given up to this point will remain part of the study, unless I ask for this to be removed in which case no data will be used. | Yes | No | |
| ☐ I understand how the researcher will use my responses, who will see them and how the data will be stored. | Yes | No | |
| ☐ I agree to take part in the above study | Yes | No | |
| Name ofparticipant | | | |
| Signature | | | |

| Date |
|--------------------|
| Name of researcher |
| taking consent |

## **Contact information of researcher**

XXXXXXXXXXXXX Programme Leader MSc Advanced Physiotherapy The University of Salford The Crescent Salford M5 4WT

0161 295 0700

XXXXXX@salford.ac.uk